CLINICAL TRIAL: NCT02135029
Title: A Phase 3, Double-blind, Double-dummy, Randomized, Placebo And Active Controlled, Parallel-group Study To Assess The Efficacy, Safety And Tolerability Of Pf-04950615 In Subjects With Dyslipidemia Who Are Intolerant To Statins
Brief Title: Randomized Clinical Trial of Bococizumab (PF-04950615; RN316) in Subjects Who Are Intolerant to Statins
Acronym: SPIRE-SI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1481030; STATIN INTOLERANT; SPIRE-SI (Other: Alias Study Number)
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-11

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia; statin intolerance
MeSH Terms: conditions — Hyperlipidemias | interventions — bococizumab; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bococizumab (PF-04950615;RN316) (Experimental): Bococizumab (PF-04950615;RN316)
  Interventions: Drug: Bococizumab (PF-04950615;RN316)
- Atorvastatin (Active Comparator)
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo for Bococizumab (PF-04950615;RN316); Other: Placebo for atorvastatin

INTERVENTIONS:
Drug: Bococizumab (PF-04950615;RN316) — 150 mg every 2 weeks by subcutaneous injection for 24 weeks
  Arms: Bococizumab (PF-04950615;RN316)
Drug: Atorvastatin — Atorvastatin PO QD
  Arms: Atorvastatin
Other: Placebo for Bococizumab (PF-04950615;RN316) — 150 mg every 2 weeks by subcutaneous injection for 24 weeks
  Arms: Placebo
Other: Placebo for atorvastatin — PO QD
  Arms: Placebo

SUMMARY:
This study is a multicenter, double blinded, active and placebo controlled randomized clinical trial to demonstrate a superior lipid lowering effect of Bococizumab (PF-04950615; RN316) compared to placebo in subjects who are statin intolerant.

ELIGIBILITY:
Inclusion Criteria:

* Hyperlipidemia
* Statin Intolerant
* Fasting LDL-C > = 70 mg/dL Fasting TG < = 400 mg/dL

Exclusion Criteria:

* Pregnant or breastfeeding females
* Cardiovascular or cerebrovascular event or procedure within 90 days
* Severe or life-threatening adverse events with past use of statins
* Poorly controlled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (31):
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Watson Clinic Center for Research, Inc. (for Drug Shipment only), Lakeland, Florida
  - Cardiovascular Research Center Of South Florida, Miami, Florida
  - St. Johns Center for Clinical Research, Ponte Vedra, Florida
  - Progressive Medical Research, Port Orange, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - NorthShore University HealthSystem - Evanston Hospital, Evanston, Illinois
  - Health Care Centers of Illinois Mokena Medical Commons, Mokena, Illinois
  - Advocate Medical Group Cardiology, Normal, Illinois
  - Advocate Medical Group Midwest Heart Specialists, Park Ridge, Illinois
  - Prairie Education & Research Cooperative (Administrative), Springfield, Illinois
  - Prairie Heart Institute, Springfield, Illinois
  - St. John's Hospital, Springfield, Illinois
  - The University of Iowa - College of Public Health - Preventive Intervention Center, Iowa City, Iowa
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Crescent City Clinical Research Center, Metairie, Louisiana
  - Allina Health System, dba Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Dayton Heart Center, Dayton, Ohio
  - Clinical and Translational Research Center, Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Berks Cardiologists, Ltd., Wyomissing, Pennsylvania
  - PMG Research of Bristol, Bristol, Tennessee
  - PMG Research of Knoxville, LLC, Knoxville, Tennessee
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Office of Michelle Zaniewski MD., PA., Houston, Texas
  - Utah Cardiology, P.C., Layton, Utah
  - Aspen Clinical Research LLC, Orem, Utah
- Canada (9):
  - The Medical Arts Health Research Group, Kelowna, British Columbia
  - Corunna Medical Research Centre, Corunna, Ontario
  - The Office of Dr. James Cha, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Devonshire Clinical Research Inc., Woodstock, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Omnispec clinical research inc., Mirabel, Quebec
  - Clinique des maladies lipidiques de Quebec, Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] Ridker PM, Tardif JC, Amarenco P, Duggan W, Glynn RJ, Jukema JW, Kastelein JJP, Kim AM, Koenig W, Nissen S, Revkin J, Rose LM, Santos RD, Schwartz PF, Shear CL, Yunis C; SPIRE Investigators. Lipid-Reduction Variability and Antidrug-Antibody Formation with Bococizumab. N Engl J Med. 2017 Apr 20;376(16):1517-1526. doi: 10.1056/NEJMoa1614062. Epub 2017 Mar 17. PMID 28304227
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481030&StudyName=Randomized%20Clinical%20Trial%20of%20RN316%20%28PF-04950615%29%20in%20Subjects%20who%20are%20Intolerant%20to%20Statins

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received single dose of placebo matched to PF-04950615 subcutaneous (SC) injection every 2 weeks along with placebo matched to Atorvastatin tablet once daily for up to 24 weeks.
- PF-04950615 150 Milligram (mg) + Placebo: Participants received single dose of PF-04950615 150 mg SC injection every 2 weeks along with placebo matched to Atorvastatin tablet once daily for up to 24 weeks.
- Atorvastatin 40 mg + Placebo: Participants received single dose of Atorvastatin 40 mg tablet once daily along with placebo matched to PF-04950615 SC injection every 2 weeks for up to 24 weeks.
Period: Overall Study
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Started | 73 | 74 | 37
Treated | 73 | 74 | 36
Completed | 69 | 69 | 34
Not Completed | 4 | 5 | 3
Not completed — Adverse Event | 2 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Other | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo | Total
Number analyzed (Participants) | 73 | 74 | 37 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (8.4) | 64 (9.2) | 65.1 (7.6) | 63.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 21 | 99
  Male | 35 | 34 | 16 | 85

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: FAS included all participants who were randomized. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent (%) change
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 70 | 71 | 35
percent (%) change | 2.4 (12.86) | -52.0 (22.75) | -32.6 (20.98)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Test type: Superiority or Other; p < 0.001, MMRM; Mixed Model Repeated Measures (MMRM); Least Square (LS) Mean Difference = -54.5, 95% CI 2-sided [-60.1 to -49.0], Standard Error of Mean 2.82 — LS-mean differences,associated 95% confidence interval (CI), and p-values were derived from an MMRM model with fixed effects for treatment group, visit,treatment group*visit interaction,baseline value, baseline value*visit*group interaction, country

2. Secondary Outcome: Percent Change From Baseline in Fasting Total Cholesterol (TC) at Weeks 12 and 24
Time Frame: Baseline, Week 12, 24
Population: FAS included all participants who were randomized. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
percent change
  Percent change at Week 12: number analyzed (Participants) | 71 | 69 | 35
  Percent change at Week 12 | 1.3 (9.92) | -37.0 (17.08) | -25.7 (16.98)
  Percent change at Week 24: number analyzed (Participants) | 70 | 68 | 33
  Percent change at Week 24 | -0.5 (11.77) | -31.2 (21.31) | -26.8 (16.64)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -38.4, 95% CI 2-sided [-42.6 to -34.2], Standard Error of Mean 2.13 — LS-mean differences, associated 95% CI, and p-values were derived from an MMRM model with fixed effects for treatment group, visit, treatment group* visit interaction, baseline value, baseline value* visit* group interaction, country
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 24; Test type: Superiority or Other; LS Mean Difference = -31.0, 95% CI 2-sided [-35.9 to -26.2], Standard Error of Mean 2.47 — LS-mean differences, associated 95% CI, for treatment group, visit, treatment group* visit interaction, baseline value, baseline value* visit* group interaction, country

3. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein B (ApoB) at Weeks 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
percent change
  Percent change at Week 12: number analyzed (Participants) | 72 | 71 | 35
  Percent change at Week 12 | 0.9 (11.64) | -46.0 (22.19) | -27.2 (18.75)
  Percent change at Week 24: number analyzed (Participants) | 70 | 70 | 33
  Percent change at Week 24 | 0.1 (13.34) | -39.1 (26.85) | -28.1 (20.20)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -46.5, 95% CI 2-sided [-51.9 to -41.1], Standard Error of Mean 2.72 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 24; Test type: Superiority or Other; LS Mean Difference = -39.3, 95% CI 2-sided [-45.4 to -33.2], Standard Error of Mean 3.10 — [estimate comment as in outcome 2, analysis 2]

4. Secondary Outcome: Percent Change From Baseline in Fasting Non High Density Lipoprotein Cholesterol (Non HDL-C) at Weeks 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
percent change
  Percent change at Week 12: number analyzed (Participants) | 70 | 69 | 35
  Percent change at Week 12 | 1.1 (11.16) | -50.0 (21.06) | -32.5 (21.24)
  Percent change at Week 24: number analyzed (Participants) | 70 | 68 | 33
  Percent change at Week 24 | -0.3 (14.46) | -41.9 (26.00) | -34.0 (21.14)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -51.2, 95% CI 2-sided [-56.3 to -46.0], Standard Error of Mean 2.61 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 24; Test type: Superiority or Other; LS Mean Difference = -41.8, 95% CI 2-sided [-47.7 to -35.8], Standard Error of Mean 3.02 — [estimate comment as in outcome 2, analysis 2]

5. Secondary Outcome: Percent Change From Baseline in Fasting Lipoprotein (a) (Lp[a]) at Weeks 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
percent change
  Percent change at Week 12: number analyzed (Participants) | 72 | 70 | 34
  Percent change at Week 12 | 2.0 (33.13) | -21.5 (39.77) | 5.1 (29.77)
  Percent change at Week 24: number analyzed (Participants) | 70 | 70 | 33
  Percent change at Week 24 | 0.8 (34.59) | -16.6 (31.71) | 4.1 (31.33)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = -23.3, 95% CI 2-sided [-35.7 to -10.8], Standard Error of Mean 6.32 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 24; Test type: Superiority or Other; LS Mean Difference = -17.4, 95% CI 2-sided [-29.6 to -5.1], Standard Error of Mean 6.21 — [estimate comment as in outcome 2, analysis 2]

6. Secondary Outcome: Percent Change From Baseline in Fasting High Density Lipoprotein Cholesterol (HDL-C) at Weeks 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
percent change
  Percent change at Week 12: number analyzed (Participants) | 70 | 70 | 35
  Percent change at Week 12 | 0.4 (12.31) | 13.2 (19.73) | 0.4 (13.51)
  Percent change at Week 24: number analyzed (Participants) | 70 | 69 | 33
  Percent change at Week 24 | -0.3 (12.34) | 11.5 (18.84) | 0.2 (14.02)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; p < 0.001, MMRM; LS Mean Difference = 12.4, 95% CI 2-sided [7.8 to 17.0], Standard Error of Mean 2.34 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 24; Test type: Superiority or Other; LS Mean Difference = 11.5, 95% CI 2-sided [6.7 to 16.4], Standard Error of Mean 2.47 — [estimate comment as in outcome 2, analysis 2]

7. Secondary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 69 | 70 | 33
percent change | 1.6 (15.62) | -42.7 (29.50) | -33.3 (20.91)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 24; Test type: Superiority or Other; LS Mean Difference = -44.8, 95% CI 2-sided [-51.3 to -38.2], Standard Error of Mean 3.33 — [estimate comment as in outcome 2, analysis 2]

8. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides (TG) at Weeks 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
percent change
  Percent change at Week 12: number analyzed (Participants) | 71 | 70 | 35
  Percent change at Week 12 | 2.2 (26.77) | -12.5 (27.42) | -20.7 (23.96)
  Percent change at Week 24: number analyzed (Participants) | 70 | 69 | 33
  Percent change at Week 24 | -3.3 (30.01) | -13.6 (40.58) | -21.9 (30.19)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; LS Mean Difference = -14.3, 95% CI 2-sided [-23.5 to -5.2], Standard Error of Mean 4.67 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 24; Test type: Superiority or Other; LS Mean Difference = -9.7, 95% CI 2-sided [-19.8 to 0.4], Standard Error of Mean 5.14 — [estimate comment as in outcome 2, analysis 2]

9. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein A-I (ApoA-I) at Weeks 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
percent change
  Percent change at Week 12: number analyzed (Participants) | 72 | 71 | 35
  Percent change at Week 12 | 1.9 (11.38) | 8.0 (14.94) | -2.8 (11.66)
  Percent change at Week 24: number analyzed (Participants) | 70 | 70 | 33
  Percent change at Week 24 | 2.3 (11.91) | 8.0 (14.66) | -2.2 (11.66)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; LS Mean Difference = 6.1, 95% CI 2-sided [2.2 to 10.1], Standard Error of Mean 2.00 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 24; Test type: Superiority or Other; LS Mean Difference = 5.6, 95% CI 2-sided [1.5 to 9.7], Standard Error of Mean 2.09 — [estimate comment as in outcome 2, analysis 2]

10. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein A-II (ApoA-II) at Weeks 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
percent change
  Percent change at Week 12: number analyzed (Participants) | 72 | 70 | 35
  Percent change at Week 12 | -0.4 (10.83) | 4.1 (13.45) | -3.2 (12.78)
  Percent change at Week 24: number analyzed (Participants) | 70 | 70 | 33
  Percent change at Week 24 | -2.2 (12.80) | 3.9 (13.21) | -0.6 (19.96)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; LS Mean Difference = 4.7, 95% CI 2-sided [0.8 to 8.7], Standard Error of Mean 2.02 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 24; Test type: Superiority or Other; LS Mean Difference = 6.5, 95% CI 2-sided [2.4 to 10.5], Standard Error of Mean 2.07 — [estimate comment as in outcome 2, analysis 2]

11. Secondary Outcome: Percent Change From Baseline in Fasting Very Low Density Lipoprotein Cholesterol (VLDL-C) at Weeks 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
percent change
  Percent change at Week 12: number analyzed (Participants) | 71 | 70 | 35
  Percent change at Week 12 | 2.2 (26.77) | -12.5 (27.42) | -20.7 (23.96)
  Percent change at Week 24: number analyzed (Participants) | 70 | 69 | 33
  Percent change at Week 24 | -3.3 (30.01) | -13.6 (40.58) | -21.9 (30.19)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; LS Mean Difference = -14.3, 95% CI 2-sided [-23.5 to -5.2], Standard Error of Mean 4.67 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 24; Test type: Superiority or Other; LS Mean Difference = -9.7, 95% CI 2-sided [-19.8 to 0.4], Standard Error of Mean 5.14 — [estimate comment as in outcome 2, analysis 2]

12. Secondary Outcome: Absolute Change From Baseline in Fasting Low Density Lipoprotein Cholesterol (LDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
milligrams per deciliter (mg/dL)
  Baseline: number analyzed (Participants) | 72 | 74 | 36
  Baseline | 182.1 (46.96) | 168.8 (47.31) | 169.9 (46.44)
  Change at Week 12: number analyzed (Participants) | 70 | 71 | 35
  Change at Week 12 | 3.1 (21.12) | -88.0 (43.82) | -56.5 (40.68)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; LS Mean Difference = -93.8, 95% CI 2-sided [-103.5 to -84.1], Standard Error of Mean 4.93 — [estimate comment as in outcome 2, analysis 2]

13. Secondary Outcome: Absolute Change From Baseline in Fasting Total Cholesterol (TC) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
mg/dL
  Baseline: number analyzed (Participants) | 73 | 72 | 36
  Baseline | 262.3 (51.20) | 250.1 (54.50) | 256.2 (53.55)
  Change at Week 12: number analyzed (Participants) | 71 | 69 | 35
  Change at Week 12 | 3.2 (25.46) | -93.8 (47.94) | -67.7 (46.85)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; LS Mean Difference = -98.7, 95% CI 2-sided [-109.9 to -87.5], Standard Error of Mean 5.67 — [estimate comment as in outcome 2, analysis 2]

14. Secondary Outcome: Absolute Change From Baseline in Fasting High Density Lipoprotein Cholesterol (HDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
mg/dL
  Baseline: number analyzed (Participants) | 73 | 73 | 36
  Baseline | 51.6 (13.92) | 51.1 (15.02) | 55.7 (13.50)
  Change at Week 12: number analyzed (Participants) | 70 | 70 | 35
  Change at Week 12 | 0.1 (6.31) | 6.0 (8.01) | -0.5 (7.07)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; LS Mean Difference = 5.9, 95% CI 2-sided [3.7 to 8.0], Standard Error of Mean 1.11 — [estimate comment as in outcome 2, analysis 2]

15. Secondary Outcome: Absolute Change From Baseline in Fasting Non High Density Lipoprotein Cholesterol (Non HDL-C) at Week 12
Time Frame: Baseline, Week 12
Population: FAS included all participants who were randomized. Here, 'n' signifies those participants who were evaluable at specified timepoint for each arm, respectively.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
mg/dL
  Baseline: number analyzed (Participants) | 73 | 72 | 36
  Baseline | 210.7 (49.75) | 199.2 (50.40) | 200.5 (50.16)
  Change at Week 12: number analyzed (Participants) | 70 | 69 | 35
  Change at Week 12 | 2.2 (22.69) | -99.8 (46.99) | -67.1 (45.59)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; LS Mean Difference = -103.6, 95% CI 2-sided [-114.6 to -92.7], Standard Error of Mean 5.56 — [estimate comment as in outcome 2, analysis 2]

16. Secondary Outcome: Absolute Change From Baseline in Fasting Triglycerides (TG) at Week 12
Time Frame: Baseline, Week 12
Population: Due to changes in planned analyses the data was not collected for this outcome measure.
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Absolute Change From Baseline in Apolipoprotein B (ApoB) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
mg/dL
  Baseline: number analyzed (Participants) | 73 | 74 | 36
  Baseline | 133.3 (27.00) | 125.8 (31.43) | 124.6 (29.82)
  Change at Week 12: number analyzed (Participants) | 72 | 71 | 35
  Change at Week 12 | 1.1 (15.08) | -57.5 (28.57) | -35.3 (25.66)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; LS Mean Difference = -59.2, 95% CI 2-sided [-66.0 to -52.4], Standard Error of Mean 3.46 — [estimate comment as in outcome 2, analysis 2]

18. Secondary Outcome: Absolute Change From Baseline in Lipoprotein (A) (Lp[A]) at Week 12
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
mg/dL
  Baseline: number analyzed (Participants) | 73 | 74 | 36
  Baseline | 32.0 (38.46) | 27.1 (36.31) | 31.7 (38.26)
  Change at Week 12: number analyzed (Participants) | 72 | 70 | 34
  Change at Week 12 | 0.7 (5.19) | -5.8 (7.93) | 1.9 (5.27)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; LS Mean Difference = -6.6, 95% CI 2-sided [-8.7 to -4.5], Standard Error of Mean 1.06 — [estimate comment as in outcome 2, analysis 2]

19. Secondary Outcome: Absolute Change From Baseline in Fasting Total Cholesterol (TC)/ High Density Lipoprotein Cholesterol (HDL-C) Ratio at Weeks 12 and 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
ratio
  Baseline: number analyzed (Participants) | 73 | 72 | 36
  Baseline | 5.4 (1.53) | 5.2 (1.45) | 4.8 (1.27)
  Absolute change at Week 12: number analyzed (Participants) | 70 | 69 | 35
  Absolute change at Week 12 | 0.1 (0.76) | -2.3 (1.13) | -1.3 (1.13)
  Absolute change at Week 24: number analyzed (Participants) | 70 | 68 | 33
  Absolute change at Week 24 | 0.0 (0.77) | -2.0 (1.35) | -1.3 (1.13)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; LS Mean Difference = -2.4, 95% CI 2-sided [-2.7 to -2.1], Standard Error of Mean 0.15 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 24; Test type: Superiority or Other; LS Mean Difference = -2.1, 95% CI 2-sided [-2.4 to -1.7], Standard Error of Mean 0.16 — [estimate comment as in outcome 2, analysis 2]

20. Secondary Outcome: Absolute Change From Baseline in Fasting Apolipoprotein B (ApoB)/Apolipoprotein A-I (ApoA-I) Ratio at Weeks 12 And 24
Time Frame: Baseline, Week 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
ratio
  Baseline: number analyzed (Participants) | 73 | 74 | 36
  Baseline | 0.9 (0.25) | 0.9 (0.24) | 0.8 (0.21)
  Absolute change at Week 12: number analyzed (Participants) | 72 | 71 | 35
  Absolute change at Week 12 | -0.0 (0.10) | -0.4 (0.21) | -0.2 (0.17)
  Absolute change at Week 24: number analyzed (Participants) | 70 | 70 | 33
  Absolute change at Week 24 | -0.0 (0.12) | -0.4 (0.25) | -0.2 (0.18)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 12; Test type: Superiority or Other; LS Mean Difference = -0.4, 95% CI 2-sided [-0.5 to -0.4], Standard Error of Mean 0.03 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 150 Milligram (mg) + Placebo; Week 24; Test type: Superiority or Other; LS Mean Difference = -0.4, 95% CI 2-sided [-0.4 to -0.3], Standard Error of Mean 0.03 — [estimate comment as in outcome 2, analysis 2]

21. Secondary Outcome: Percentage of Participants Achieving Fasting Low Density Lipoprotein Cholesterol (LDL-C) Less Than or Equal to (<=) 100 Milligram Per Deciliter (mg/dL) at Weeks 12 and 24
Time Frame: Week 12, 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
percentage of participants
  Week 12: number analyzed (Participants) | 71 | 71 | 35
  Week 12 | 1.4 | 71.8 | 42.9
  Week 24: number analyzed (Participants) | 70 | 70 | 33
  Week 24 | 0 | 61.4 | 45.5

22. Secondary Outcome: Percentage of Participants Achieving Fasting Low Density Lipoprotein Cholesterol (LDL-C) Less Than or Equal to (<=) 70 Milligram Per Deciliter (mg/dL) at Weeks 12 and 24
Time Frame: Week 12, 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 37
percentage of participants
  Week 12: number analyzed (Participants) | 71 | 71 | 35
  Week 12 | 0 | 45.1 | 14.3
  Week 24: number analyzed (Participants) | 70 | 70 | 33
  Week 24 | 0 | 41.4 | 15.2

23. Secondary Outcome: Plasma PF-04950615 Concentrations at Weeks 12 and 24
Description: Concentration versus time summary was calculated by setting concentration values below the lower limit of quantification (LLOQ =0.4 micrograms per milliliter [mcg/mL]) to zero. Participants who received PF-04950615 150 mg were evaluable for this outcome measure.
Time Frame: Week 12 and 24
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Here, 'N' signifies those participants who were evaluable for this outcome measure and 'n' signifies those participants who were evaluable at specified time point for the arm.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | PF-04950615 150 Milligram (mg) + Placebo
Number analyzed (Participants) | 72
mcg/mL
  Week 12: number analyzed (Participants) | 71
  Week 12 | 10.21 (9.309)
  Week 24: number analyzed (Participants) | 69
  Week 24 | 7.38 (7.890)

24. Secondary Outcome: Number of Participants With Adverse Events Related to Type 1 and 3 Hypersensitivity Reactions, Injection Site Reactions, Myalgia, Myopathy, Creatinine Kinase (CK) and Liver Function Tests (LFT) Elevations
Time Frame: Baseline (Day 1) up to Week 30
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 36
participants
  Type 1 and 3 hypersensitivity reactions | 1 | 0 | 0
  Injection site reactions | 4 | 16 | 0
  Myalgia | 13 | 13 | 7
  Myopathy | 0 | 0 | 0
  CK Elevations | 0 | 1 | 0
  LFT Elevations | 1 | 2 | 1

25. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) and Neutralizing Antibodies (nAb)
Description: Participants with at least one positive ADA titer greater than or equal to (>=) 6.23 or positive nAb titer >=4.32 were reported. Titers are expressed as log2 reciprocal dilution at assay cutpoint.
Time Frame: Baseline up to Week 30
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Here, 'N' signifies those participants who were evaluable for this outcome measure. Participants who received PF-04950615 150 mg were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | PF-04950615 150 Milligram (mg) + Placebo
Number analyzed (Participants) | 72
participants
  ADA | 35
  nAb | 21

26. Secondary Outcome: Anti-drug Antibody (ADA) and Neutralizing Anti-body (nAb) Titer Level in Participants Who Tested Positive for ADA and nAb Respectively
Description: Titer levels of participants who tested positive for ADA and nAb are reported. Titers are expressed as log2 reciprocal dilution at assay cutpoint.
Time Frame: Week 4, 12, 24 and 30 (Follow-up)
Population: Safety analysis set: all participants who received at least 1 dose of study treatment. Here, 'N' signifies those participants who were evaluable for this outcome measure and 'n' signifies those participants who were evaluable at specified time point for the arm. Participants who received PF-04950615 150 mg were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | PF-04950615 150 Milligram (mg) + Placebo
Number analyzed (Participants) | 35
titer
  ADA Titer: Week 4: number analyzed (Participants) | 2
  ADA Titer: Week 4 | 9.94 (1.181)
  ADA Titer: Week 12: number analyzed (Participants) | 10
  ADA Titer: Week 12 | 9.49 (1.646)
  ADA Titer: Week 24: number analyzed (Participants) | 23
  ADA Titer: Week 24 | 9.46 (2.196)
  ADA Titer: Week 30: number analyzed (Participants) | 32
  ADA Titer: Week 30 | 10.12 (2.981)
  nAb Titer: Week 4: number analyzed (Participants) | 0
  nAb Titer: Week 12: number analyzed (Participants) | 2
  nAb Titer: Week 12 | 6.05 (2.440)
  nAb Titer: Week 24: number analyzed (Participants) | 5
  nAb Titer: Week 24 | 5.28 (1.358)
  nAb Titer: Week 30: number analyzed (Participants) | 19
  nAb Titer: Week 30 | 6.09 (2.135)

27. Secondary Outcome: Percentage of Participants Discontinued Due to Myalgia, Myopathy, Creatinine Kinase (CK) and Liver Function Tests (LFT) Elevations
Time Frame: Baseline (Day 1) up to Week 30
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Number analyzed (Participants) | 73 | 74 | 36
percentage of participants
  Myalgia | 9.6 (0.10) | 10.8 (0.21) | 16.7 (0.17)
  Myopathy | 0 (0.12) | 0 (0.25) | 0 (0.18)
  CK Elevations | 0 | 0 | 0
  LFT Elevations | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | PF-04950615 150 Milligram (mg) + Placebo | Atorvastatin 40 mg + Placebo
Serious Adverse Events (participants affected / at risk) | 7/73 | 8/74 | 1/36
Other Adverse Events (participants affected / at risk) | 44/73 | 41/74 | 20/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | PF-04950615 150 Milligram (mg) + Placebo (N=74) | Atorvastatin 40 mg + Placebo (N=36)
Angina pectoris (Cardiac disorders) | 2 | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Bursitis infective (Infections and infestations) | 1 | 0 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=73) | PF-04950615 150 Milligram (mg) + Placebo (N=74) | Atorvastatin 40 mg + Placebo (N=36)
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 1
Nausea (Gastrointestinal disorders) | 2 | 4 | 2
Fatigue (General disorders) | 6 | 3 | 4
Injection site reaction (General disorders) | 2 | 14 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 2/38 | 0/40 | 0/21 — This adverse event was assessed only in female participants.
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 7 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 13 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 4 | 1
Dizziness (Nervous system disorders) | 3 | 2 | 3
Headache (Nervous system disorders) | 2 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.